CLINICAL TRIAL: NCT03178617
Title: Improving Learning and School Functioning in Latino Children With Cancer
Brief Title: High-Intensity Parent Intervention Program in Improving Learning and School Functioning in Latino Children With Acute Leukemia or Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17139; NCI-2017-00971 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17139 (Other: City of Hope Medical Center); RSG-17-023-01-CPPB (Other Grant/Funding Number: ACS)
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Lymphoblastic Lymphoma; Acute Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care LIP) (Active Comparator): Parents or caregivers attend standard of care LIP consisting of a meeting to review results of a neurocognitive evaluation and to discuss recommendations for optimal learning and school performance for 1 session.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (HIP) (Experimental): Parents or caregivers attend HIP consisting of individual parental skill training sessions with a bilingual therapist over 60-90 minutes every 2 weeks for a total of 8 sessions.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend standard of care LIP
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (standard of care LIP)
Other: Educational Intervention — Attend HIP
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (HIP)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well a high-intensity intervention parenting program works in improving learning and school functioning in Latino children with acute leukemia or lymphoblastic lymphoma. A high-intensity intervention program may help doctors to see whether training parents or caregivers in specific parenting skills and "pro-learning" behaviors will result in better learning and school outcomes for Latino children with acute leukemia or lymphoblastic lymphoma. It is not yet known if a high-intensity intervention program is more beneficial than a standard of care lower intensity parenting intervention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effectiveness of an enhanced parenting intervention, high-intensity intervention program (HIP), on pediatric cancer survivors' learning and school health-related quality of life (HRQOL) outcomes up to 12 months post enrollment.

II. Determine the effectiveness of HIP on the "pro-learning" efficacy of parents of pediatric cancer survivors up to 12 months post enrollment.

III. Examine the extent to which the parent's increases in personal efficacy and use of "pro-learning" behaviors correlate with the child's school HRQOL and academic performance.

IV. Obtain preliminary data on the relationships between family stress and the Val66Met polymorphism of brain-derived neurotrophic factor (BDNF) with neurocognitive and health-related quality of life (HRQOL) outcomes in Latino children treated with CNS-directed therapies for cancer.

V. Conduct preliminary analysis on the interaction between family stress and the BDNF Met polymorphism when predicting cognitive and HRQOL outcomes in Latino children treated for cancer.

EXPLORATORY OBJECTIVES:

I. Explore the associations between neurocognitive performance and polymorphisms in candidate genes previously reported to explain cognitive variability in childhood cancer survivors (e.g., the catechol-O-methyltransferase Val158Met polymorphism and the nitric oxide synthase [NOS3] 894T allele) or involved in the stress response (e.g., the Serotonin transporter rs25531 and the Glucocorticoid receptor rs6190).

OUTLINE: Parents or caregivers are randomized to 1 of 2 arms.

ARM I: Parents or caregivers attend standard of care lower intensity intervention program (LIP) consisting of a meeting to review results of a neurocognitive evaluation and to discuss recommendations for optimal learning and school performance for 1 session.

ARM II: Parents or caregivers attend HIP consisting of individual parental skill training sessions with a bilingual therapist over 60-90 minutes every 2 weeks for a total of 8 sessions.

After study enrollment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PARENT/CAREGIVER: Adult primary caregiver of children treated for leukemia or lymphoblastic lymphoma (LL) and daily contact with the child
* PARENT/CAREGIVER: One or both parents self-identify as Hispanic/Latino and the primary participating parent/caregiver is monolingual or bilingual Spanish speaking
* CHILD: Children treated for acute leukemia (e.g. acute lymphoblastic leukemia [ALL], acute myeloid leukemia [AML]), LL, or other types of leukemia (if treated intensively) aged 5-12 years and their parents/caregivers
* CHILD: Child has completed cancer treatment and is up to 10 years post-treatment
* CHILD: Child understands English and is enrolled in school (but can be bilingual)

Exclusion Criteria:

* History of major psychiatric condition (e.g. psychosis) in parent or child; severe neurodevelopmental disorder in child (e.g. Down's syndrome)
* Recent or current participation in educational/behavioral intervention study with similar focus

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Change in child's health-related quality of life school functioning | Baseline up to 12 months
  Measured by the parent-reported Pediatric Quality of Life Inventory school domain.
Change in parental efficacy | Baseline up to 12 months
  Measured by the Efficacy scale from the Parent Knowledge, Beliefs and Behaviors Questionnaire-3rd Revision (PBQ-R3).

SECONDARY OUTCOMES:
Objective academic performance (Child) | Up to 12 months
  Measured by WIAT: reading and math scores and classroom grades from school report cards.
Attention performance (Child) | Up to 12 months
  Measured by the Conners Parent Report Attention subscale.
Frequency of pro-learning behaviors (Parent) | Up to 12 months
  Measured by PBQ-R3 Behaviors Scale.
Frequency of pro-learning behaviors (Parent) | Up to 12 months
  Measured by the Parents' weekly time spent with child in pro-learning behaviors and activities.
Knowledge of pro-learning parenting (Parent) | Up to 12 months
  Measured by PBQ-R3 Knowledge scale.
Children's scores on other neurocognitive tests as assessed by learning, memory, and processing speed | Up to 12 months
Parental reports of their children's HRQOL as measured by the PedsQL parent proxy questionnaire | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Patel, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California